CLINICAL TRIAL: NCT00494273
Title: HIV Prevention in Haitian Youths (HAP)
Brief Title: HIV Prevention in Haitian American Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD038458 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: Haitian American Adolescents; HIV Prevention; Cognitive Behavioral Intervention
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral and Standard Care with Healthy Living

SUMMARY:
There has not been a great deal of research involving Haitian American adolescents and HIV risk reduction. The purpose of the study is to learn better ways to teach teenagers about living healthy by educating these children about how to make good choices about things like eating healthy, exercise, and sexual behavior. The primary focus of the proposed study is to understand the mechanisms of adopting safer sex practices among Haitian American (H-A) adolescents. We will enroll 160 male and 160 female participants to achieve the target sample of 272 participants at the 12-month follow-up time point.

DETAILED DESCRIPTION:
The primary focus of the study is to understand the mechanisms of adopting safer sex practices among Haitian American (H-A) adolescents. We replicated a Cognitive-Behavioral HIV transmission risk reduction (CB-HIV-TRR) intervention entitled "Becoming A Responsible Teen" (BART, St. Lawrence, et al, 1995; St. Lawrence, 1998). This approach, which emphasizes building skills and self-efficacy in the process of risk reduction, was demonstrated to be highly effective with African American male and female adolescents in Mississippi. In a meta-analysis of published CB-HIV-RR intervention outcome studies (Kalichman, et al., 1996), the BART intervention was shown to have produced the highest effect not only for the published studies with adolescents, but also for HIV prevention interventions of all other populations studied. Based on its promising effects, the BART intervention has been officially designed as one of only four HIV risk "Programs that Work" by CDC Division of Adolescent and School Health (DASH). CDC designates programs as such based on reviewing programs in the literature using rigorous criteria. The proposed work focused on delineating theoretically important conditions associated with HIV transmission risk reduction (HIV-TRR) to address issues of mechanism of action and generalizability, respectively. Specifically, this 5 year study evaluates the effects of a version of the BART intervention that has been adapted to be appropriate to Haitian adolescents in Miami) as compared to a standard care (SC) condition among 160 male and 160 female high risk Haitian adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. The adolescent reports being at high risk for HIV transmission by virtue of having ever engaged in risky sexual behavior.
2. The adolescent is available for the full duration of the study with no anticipated circumstances impeding study participation (e.g., jail term, out-of-town, etc.).
3. The adolescent is fluent in spoken English required to complete our assessment battery and participate in group interventions. Because all of the adolescent are in or have been in the English speaking Public School system they virtually all are fluent in English.
4. The adolescent is willing to assent for participation in the study.
5. The adolescent has an identifiable parent or parent-figure (i.e., a number of adolescents will have sisters, aunts, or grandmothers who function as their primary caretaker) who is the legal guardian for the adolescent and who is willing to sign the informed consent. A bilingual assessor who is fluent in Creole will be available to parents that speak limited English and the consent forms for the parents will be in Creole.
6. The adolescent is assessed not to be harmful to self or others using the relevant sections of the POSIT-HRS and Millon Adolescent Clinical Inventory (MACI).
7. The adolescent has no evidence of psychiatric impairments (e.g., psychosis) that might compromise the participants' ability to comprehend and participate in the assessment and intervention processes.
8. The child's guardian will be invited to complete a questionnaire regarding communication with their teenager about sex and their guardian's level of acculturation.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320
Dates: Start 2002-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The BART Condition will reduce HIV transmission risk behavior over time more than the SC. Assessments will be completed prior, after, 4 , 8 and 12 months after the intervention. Measure examples are
Sexual and Condom Attitudes
Self-Efficacy Scale
Behavioral Intentions scale
Health Protective Sexual Communication Scale
Comfort talking about Safer Sex measure
Condom Use Skills
Risk Behavior Assessment

SECONDARY OUTCOMES:
Examples are
The Millon Adolescent Clinical Inventory
The Adolescent-Family Inventory of Life Events & Changes
Stephenson Multigroup Acculturation Scale
Adolescent Health Questionnaire-Adolescent and Parent Version.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Malow, Ph.D., Principal Investigator — Florida International University
Locations (1):
- Center for Haitian Studies, Miami, Florida, United States